CLINICAL TRIAL: NCT05318690
Title: PlayGait: A Dynamic Exoskeleton to Improve Community Ambulation
Brief Title: PlayGait: A Dynamic Exoskeleton
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty with recruitment
Sponsor: Orthocare Innovations, LLC (Industry)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: 0047-01
Record Dates: First submitted 2022-03-24; First posted 2022-04-08 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Cerebral Palsy
Keywords: pediatric; orthosis; exoskeleton
MeSH Terms: conditions — Cerebral Palsy | interventions — BaseLine dental cement

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PlayGait (Exoskeleton) (Experimental): Experimental lower-limb device.
  Interventions: Device: PlayGait
- Baseline (Active Comparator): Baseline condition without using any prescribed lower-limb orthoses.
  Interventions: Other: Baseline

INTERVENTIONS:
Device: PlayGait — PlayGait is a dynamic energy storing and returning lower-limb exoskeleton.
  Arms: PlayGait (Exoskeleton)
Other: Baseline — Baseline condition with no prescribed or intervention lower-limb devices.
  Arms: Baseline

SUMMARY:
PlayGait is an investigational dynamic energy storage and return (ESR) lower-limb exoskeleton for young children with cerebral palsy (CP), that stores energy while the child is in the stance phase of walking and returns that energy in terminal stance and early swing phase of walking. PlayGait assists with the passive dynamics of walking through an exotendon (comprised of a spring in series with a cable). The overall objective of this investigational device is to promote correct walking patterns that encourage proper bone alignment, muscle recruitment, and strengthening during walking practice in young children with CP. The study will evaluate children with CP's activity levels in the community with and without PlayGait. The study will consist of three lab visits and two, 7-day periods at home.

ELIGIBILITY:
Inclusion Criteria:

* Age 3 - 4 years (at time of informed consent)
* Hemiplegic cerebral palsy
* If child uses an ankle-foot orthosis (AFO), parent/caregiver is willing to have the child stop wearing their prescribed AFO during data collections (lab sessions and two 7-day periods at home)
* Ability to walk at least 10 meters without the use of assistive devices or AFOs
* Ability to walk at least 1 minute without the use of assistive devices or AFOs
* Stiff knee gait - less than normal knee flexion during swing phase
* Hip flexion passive range of motion contracture less than 20 degrees
* Gross Motor Function Classification System (GMFCS) Levels I-II
* Modified Ashworth Scale (MAS) <=2 for the gastrocnemius soleus, rectus femoris, and hamstrings
* Family has resources to attend all study sessions (transportation, schedule)
* Ability to speak and understand in English

Exclusion Criteria:

* Orthopedic surgery in the last year
* Foster children or wards of the state
* Use wheelchair or stroller mobility as their primary method of independent mobility
* Severe visual impairment such that the visual impairment itself functionally limits mobility
* Phenol or Botox injections to the legs in the last 3 months
* Uncontrolled seizure disorder, defined as any seizure in the last 3 months that influenced mobility skills and function (seizures which did not affect mobility are acceptable)
* Lower limb fracture in the last 3 months
* Planned surgery or changes to movement disorder medication during the study period
* Inability to understand directions sufficiently to complete the study assessments
* Cognitive, behavioral, or any other issues that may not allow for effective study participation
* Unwilling to complete the study protocol

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-01-03 (Actual)

PRIMARY OUTCOMES:
Cadence | 7 days with baseline condition; 7 days with PlayGait condition
  Low, medium, and high activity rate
Shifts in cadence | 7 days with baseline condition; 7 days with PlayGait condition
  Shifts from low to medium cadence and shifts from medium to high cadence

SECONDARY OUTCOMES:
1 minute walk test | 1st lab session (baseline); 3rd lab session with PlayGait after 7 days of wearing PlayGait
  The distance walked in one minute
10 meter walk test | 1st lab session (baseline); 3rd lab session with PlayGait after 7 days of wearing PlayGait
  The time it takes to walk 10 meters
Pediatric Balance Scale | 1st lab session (baseline); 3rd lab session with PlayGait after 7 days of wearing PlayGait
  Participant completes 14 activity items that measure pediatric balance
Average steps per day | Baseline Condition: 7 days in the community without PlayGait (no lower-limb assistive devices); PlayGait condition: 7 days with PlayGait
  Step count per day
Time of PlayGait use | PlayGait condition: 7 days in the community with PlayGait
  Amount of time each day that PlayGait is worn

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Zistatsis, MSME, Principal Investigator — Orthocare Innovations
Locations (1):
- Orthocare Innovations, LLC, Edmonds, Washington, United States